CLINICAL TRIAL: NCT03934229
Title: The Effect of the Probiotic Bifidobacterium Animalis Ssp. Lactis 420 (B420) on Body Fat Mass in Overweight and Obese Individuals Following Healthy Lifestyle Intervention: A Randomized, Double-blind, Placebo-controlled, Multi-center Study
Brief Title: Effect of Study Probiotics on Body Fat Mass in Overweight and Obese Individuals Following Healthy Lifestyle Intervention
Acronym: QLSlimCapHL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danisco France SAS (Industry)
Collaborators: Eurofins Optimed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2018-A03140-55
Record Dates: First submitted 2019-04-18; First posted 2019-05-01 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Overweight; Obesity
Keywords: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Active (Experimental): Bifidobacterium animalis ssp. lactis 420 at 1*10^10 colony forming units (CFU) per day
  Interventions: Dietary Supplement: Daily intake of study product
- Group Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Daily intake of study product

INTERVENTIONS:
Dietary Supplement: Daily intake of study product — Daily intake of Bifidobacterium animalis ssp. lactis 420 or placebo for a 6-month period

SUMMARY:
A randomized, double-blind, placebo-controlled, multi-center, parallel group study on overweight and obese individuals following healthy lifestyle consisting of calorie-reduced diet (20% calorie restriction) and increase in daily activity (1000 steps more per day once compared to the baseline steps)

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary, written, signed, informed consent to participate in the study
2. Male or female, age between 20 to 65 (inclusive)
3. BMI between 28.0 and 34.9 (inclusive), of which 1:1 overweight (28.0-29.9):obese (30-34.9)
4. Waist circumference for men of > 102 cm or for women of > 88 cm
5. Agreement to comply with the protocol and study restrictions
6. Access to Internet in addition to willingness and ability to use web-based questionnaires
7. Available for all study visits
8. Females of child-bearing potential required to provide a negative urine pregnancy test and agree to use a medically-approved method of birth control, eg. all of the following are approved: birth control pill, patch, shot, vaginal ring, mini pill, long-acting reversible contraception (LARC) meaning hormonal intrauterine device, nonhormonal intrauterine device with copper, subdermal contraceptive implant, condoms, cervical cap, diaphragm.
9. Covered by Health Insurance System and / or in compliance with the recommendations of National Law in force relating to biomedical research.

Exclusion Criteria:

1. Diagnosed and pharmacologically-treated type 1 and type 2 diabetes (fasting blood glucose ≥ 7 mmol/l)
2. Use of medication/supplements for blood glucose control
3. Pharmacologically-treated (medication/supplements) hypertension or dyslipidemia
4. Cardiovascular disease, hypertensive retinopathy, left ventricular dysfunction, secondary hypertension, liver dysfunction/disease, kidney dysfunction/disease, dementia, thyroid disease, pancreatic disease, history of cancer within past 5 years (excluding basal cell carcinoma), anemia, or any other disease or condition which, in the Investigator's opinion, could interfere with the results of the study or the safety of the subject
5. Use of drugs or supplements to manage body weight or body fat in the last 3 months
6. Use of laxatives or fiber supplements in the past 6 weeks.
7. History of chronic active inflammatory disorders
8. History of bariatric surgery
9. History of any chronic gastrointestinal disease (e.g. IBD) or disorders (e.g. IBS, constipation, diarrhea), or gastrointestinal reflux disease
10. Regular use of non-steroidal anti-inflammatory drugs, systemic or inhaled corticosteroids, or systemic immunomodulatory drugs
11. Regular (more than once per week) use of proton pump inhibitors
12. Recent (last 3 months) or ongoing antibiotic use
13. Immunosuppression or ongoing therapy causing immunosuppression
14. Use of probiotic supplements during the previous 6 weeks
15. Significant change in tobacco, snuff, nicotine and e-cigarette use habits in the past 3 months or planned cessation of the use of these products during the trial
16. Use of vitamin D supplementation of ≥100 µg/day
17. Active or recent (last 3 months) participation in a weight loss program (diet and/or exercise)
18. Weight change (increase or loss) of 3 kg during the past 3 months
19. Pregnant or planning pregnancy during the study or breastfeeding
20. Participation in a clinical trial with an investigational product or drug within 60 days prior to screening
21. Likeliness to be noncompliant with the protocol
22. No possibility of contact in case of emergency
23. Illicit drug users
24. Alcohol abusers
25. Administrative or legal supervision
26. Subject who would receive more than 4500 euros as indemnities for his participation in biomedical research within the 12 last months, including the indemnities for the present study
27. Other reasons that, in the opinion of the Investigator, make the participant unsuitable for enrolment
28. Other reasons that, in the opinion of the Investigator, make the participant unsuitable for enrolment

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
Total body fat mass relative change | Change from baseline at 6 months
  Difference in total body fat mass relative change from baseline (Visit 2) to 6 months of product intake (Visit 5) between the active vs. placebo group

SECONDARY OUTCOMES:
Trunk fat mass change | Change from baseline at 2 months, 4 months and 6 months
  Change in trunk fat mass from baseline (Visit 2) to 2 months (Visit 3), 4 months (Visit 4) and 6 months (Visit 5) (absolute and relative)
Waist circumference change | Change from baseline (Visit 2) to 2 months (Visit 3), 4 months (Visit 4) and 6 months (Visit 5)
  Change in waist circumference from baseline (Visit 2) to 2 months (Visit 3), 4 months (Visit 4) and 6 months (Visit 5) (absolute and relative)
Android fat mass change | Change from baseline (Visit 2) to 2 months (Visit 3), 4 months (Visit 4) and 6 months (Visit 5)
  Change in android fat mass from baseline (Visit 2) to 2 months (Visit 3), 4 months (Visit 4) and 6 months (Visit 5) (absolute and relative)
Lean body mass change | Change from baseline (Visit 2) to 2 months (Visit 3), 4 months (Visit 4) and 6 months (Visit 5)
  Change in lean body mass from baseline (Visit 2) to 2 months (Visit 3), 4 months (Visit 4) and 6 months (Visit 5) (absolute and relative)
Energy intake change | Change from baseline at 6 months
  Change in energy intake from baseline (Visit 2) to 6 months (Visit 5)
Fat mass change in individual body regions | Change from baseline (Visit 2) to 2 months (Visit 3), 4 months (Visit 4) and 6 months (Visit 5)
  Change in fat mass in other individual body regions from baseline (Visit 2) to 2 months (Visit 3), 4 months (Visit 4) and 6 months (Visit 5) (absolute and relative)
Total fat mass absolute change | Change from baseline (Visit 2) to 2 months (Visit 3), 4 months (Visit 4) and 6 months (Visit 5)
  Change in total body fat mass absolute change from baseline (Visit 2) to 2 months (Visit 3), 4 months (Visit 4) and 6 months (Visit 5)
Body weight change | Change from baseline (Visit 2) to 2 months (Visit 3), 4 months (Visit 4) and 6 months (Visit 5)
  Change in body weight from baseline (Visit 2) to 2 months (Visit 3), 4 months (Visit 4) and 6 months (Visit 5) (absolute and relative)
BMI change | Change from baseline at 6 months
  Change in BMI from baseline (Visit 2) to 6 months (Visit 5) (absolute and relative)
Hip circumference change | Change from baseline (Visit 2) to 2 months (Visit 3), 4 months (Visit 4) and 6 months (Visit 5)
  Change in hip circumference from baseline (Visit 2) to, 2 months (Visit 3), 4 months (Visit 4) and 6 months (Visit 5) (absolute and relative)
Total fat mass relative change | Change from baseline (Visit 2) to 2 months (Visit 3), and 4 months (Visit 4)
  Change in total body fat mass relative change from baseline (Visit 2) to 2 months (Visit 3), and 4 months (Visit 4)

OTHER OUTCOMES:
Food intake change | Change from baseline (Visit 2) to 2 months (Visit 3), 4 months (Visit 4) and 6 months (Visit 5)
  Change in food intake from baseline (Visit 2) to 2 months (Visit 3), 4 months (Visit 4) and 6 months (Visit 5)
Physical activity change | Change from baseline at 6 months
  Change in physical activity (IPAQ) from baseline (Visit 2) to 6 months (Visit 5)
Daily activity change | Change from baseline (Visit 2) to 2 months (Visit 3), 4 months (Visit 4) and 6 months (Visit 5)
  Change in daily activity (steps, pedometer/accelerometer) from baseline (Visit 2) to 2 months (Visit 3), 4 months (Visit 4) and 6 months (Visit 5)
Fasting glucose levels change | Change from baseline at 6 months
  Change in fasting glucose levels from baseline (Visit 2) to 6 months (Visit 5)
Fasting insulin levels change | Change from baseline at 6 months
  Change in fasting insulin levels from baseline (Visit 2) to 6 months (Visit 5)
Insulin resistance change | Change from baseline at 6 months
  Change in insulin resistance from baseline (Visit 2) to 6 months (Visit 5)
HbA1c change | Change from baseline at 6 months
  Change in glycated hemoglobin HbA1c from baseline (Visit 2) to 6 months (Visit 5)
Blood lipids change | Change from baseline at 6 months
  Change in blood lipids from baseline (Visit 2) to 6 months (Visit 5)
Inflammation markers change | Change from baseline at 6 months
  Change in inflammation markers, as specified in Section 4.2.8, from baseline (Visit 2) to 6 months (Visit 5)
Circulating zonulin change | Change from baseline at 6 months
  Change in circulating zonulin from baseline (Visit 2) to 6 months (Visit 5)
Barrier function and endotoxemia markers change | Change from baseline at 6 months
  Change in markers of gut barrier function and endotoxemia, as specified in Section 4.2.8, from baseline (Visit 2) to 6 months (Visit 5)
Fecal microbiota change | Change from baseline at 6 months
  Change in fecal microbiota from baseline (Visit 2) to 6 months (Visit 5)
Fecal metabolites change | Change from baseline at 6 months
  Change in fecal metabolites from baseline (Visit 2) to 6 months (Visit 5)
Adipose tissue biomarkers change | Change from baseline at 6 months
  Change in adipose tissue biomarkers, as specified in Section 4.2.8, from baseline (Visit 2) to 6 months (Visit 5)

CONTACTS AND LOCATIONS:
Locations (7):
- France (3):
  - CEN nutriment, Dijon
  - Eurofins Optimed, Gières
  - Biofortis SAS, Saint-Herblain
- Spain (4):
  - Cap Vallcarca, Barcelona
  - CAP Centelles, Barcelona
  - CAP Hostalets, Barcelona
  - CAP Muralles, Tarragona